CLINICAL TRIAL: NCT04592133
Title: Prospective Evaluation of Temporomandibular Joint Pathologies in Scoliosis Patients With Ultrasonography and Clinical Examination
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Merve Yelken Kendirci, Researcher, Istanbul University
Other Study IDs: 2020/1
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Scoliosis Patients
Keywords: Ultrasonography
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Scoliosis Patients
  Interventions: Diagnostic Test: Ultrasonography
- Control Group
  Interventions: Diagnostic Test: Ultrasonography

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Ultrasonography Examination

SUMMARY:
From the anatomical and functional point of view, stomatognathic system and spine have close connections. Together with the complex neuromuscular relationships, this creates an important area of cooperation between dentists and orthopedics (1). The cause of scoliosis has not been precisely explained, and various causes have been suggested in the literature, such as deviation from the standard growth pattern, neuromuscular tissue changes, asymmetric growth of the trunk, changes in the sagittal configuration of the spine, and environmental factors. In addition, scoliosis may develop secondary to each of hereditary musculoskeletal disorders such as osteogenesis imperfecta, Marfan syndrome, Stickler syndrome, Ehlers-Danlos syndrome and muscular dystrophies.

Fonder et al. conducted case studies showing the relationship between dental occlusion and scoliosis (2). There are studies suggesting that temporomandibular joint (TMJ) diseases are observed more frequently with the effect of the head-neck muscle balance affected by scoliosis and the irregularities in the occlusion. At the same time, some studies have shown that patients with mandible changes (deviation, deflection, asymmetry…), which is one of the TMJ components, often have abnormal morphology in the cervical vertebrae (3). Ito G et al. They reported that body posture is closely related to the function of the head support system. The cervical spine and muscles play an important role in stabilizing the head posture and in the complex and various movements of the head (4).

There is no study in the literature comparing the severity of scoliosis and TMJ joint dysfunction radiologically and clinically.

In this study, TMJ of scoliosis patients was evaluated by ultrasonography and clinical examination; It was aimed to correlate the severity of scoliosis with joint dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 12-18
* Being diagnosed with Adolescent Idiopathic Scoliosis

Exclusion Criteria:

* Being diagnosed with neuromuscular, juvenile or congenital scoliosis
* Having received surgical treatment for scoliosis
* Rheumatological disease
* Having received treatment for TMJ dysfunction

Ages: 12 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All patient population admitted to our clinic
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-03 (Actual); Study Completion 2021-01-03 (Actual)

PRIMARY OUTCOMES:
Joint Pain Scale | 7 month
  Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) form will be used in our study

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Dentistry Faculty, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Not

REFERENCES:
- [Background] Saccucci M, Tettamanti L, Mummolo S, Polimeni A, Festa F, Tecco S. Scoliosis and dental occlusion: a review of the literature. Scoliosis. 2011 Jul 29;6:15. doi: 10.1186/1748-7161-6-15. PMID 21801357
- [Background] Tecco S, Festa F. Cervical spine curvature and craniofacial morphology in an adult Caucasian group: a multiple regression analysis. Eur J Orthod. 2007 Apr;29(2):204-9. doi: 10.1093/ejo/cjl061. Epub 2007 Jan 11. PMID 17218718
- [Background] Ito, G., & Yamazaki, K. (1995). Relation between posture and the maxillofacial cranium. Jpn Dent Assoc, 48, 15-26.
- See also: Joint, J. (2010). TMJ. Association. TMJ diseases and disorders: Basics-overview. — http://www.tmj.org/